CLINICAL TRIAL: NCT03266042
Title: Collection of Safety, Efficacy and Resource Utilization Information in Patients Who Have Received Melphalan PHP With the Delcath Hepatic Delivery System for the Treatment of Unresectable Hepatic Malignancy
Brief Title: Registry Protocol- Melphalan Percutaneous Hepatic Perfusion for the Treatment of Unresectable Hepatic Malignancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PHP-M-REG01
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Hepatic Malignant Neoplasm Primary Non-Resectable

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Collection of Safety, Efficacy and Resource Utilization Information in Patients Who Have Received Melphalan PHP with the Delcath Hepatic Delivery System for the Treatment of Unresectable Hepatic Malignancy

DETAILED DESCRIPTION:
Post Marketing study:

The CHEMOSAT kit containing Gen 2 filters has been used to treat patients since April 2012. This registry study is designed to collect safety, resource utilization and treatment outcomes in patients who receive this treatment with CHEMOSAT by healthcare professionals. The safety and efficacy data from patients treated with CHEMOSAT is important in updating the safety profile and for collection of treatment information. The resource utilization information is essential in planning treatment strategy for patients.

This registry does not follow any pre-determined protocol with respect to diagnosis, treatment or follow-up of the patient. The data collected will be gathered exclusively from current medical practice at participating institutions.

Delcath holds a list of authorized customer hospitals to whom it supplies the CHEMOSAT System. To date these hospitals have treated over 300 patients with cancers of the liver.

The decision to treat with CHEMOSAT is clearly separated from the decision to collect data in the registry. No specific procedures or tests are required in this protocol.

ELIGIBILITY:
1. Have received CHEMOSAT treatment per IFU within the last 6-months or are planned to receive treatment with CHEMOSAT.
2. Have provided written informed consent according to institutional and regulatory guidelines

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Collection of Safety, Efficacy and Resource Utilization Information in Patients Who Have Received or will receive treatment with CHEMOSAT for the Treatment of Unresectable Hepatic Malignancy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01-14 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Gather key safety data on the use of CHEMOSAT Kit (Gen 2 filter). | Post-procedure (up to 30 days after CS-PHP)
  Data to be collected at: Baseline, treatment and post treatment laboratory values and clinical measurements until time of discharge

SECONDARY OUTCOMES:
Percentage of treatment with CHEMOSAT each patient receives | From the first CHEMOSAT treatment through the last, [timeframe an average of 12-months if 6 cycles completed]
  The percentage of treatments with CHEMOSAT each patient receives based on primary tumor
Evaluation of Best Overall Response | from the date of first CHEMOSAT treatment through last CHEMOSAT treatment, or treatment discontinuation or death (whichever occurs first) [assessed up to 24 months]
  Evaluation of patient best overall response (partial response or complete response, when applicable)
Evaluation of resource utilization | From the first CHEMOSAT treatment through the last CHEMOSAT treatment [assessed up to 24 months]
  Percentage of days spent in ICU, step-down area
Evaluate time to treatment failure | time from first CHEMOSAT treatment to the date of last CHEMOSAT treatment [assesed up to 24 months]
  Time of first CHEMOSAT treatment to time of treatment failure

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Southampton University Hospitals and University of Southampton, Southampton
  - Spire Southampton Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided